CLINICAL TRIAL: NCT02212730
Title: A Clinical Trial to Evaluate the Effect of Neoadjuvant MK-3475 (Pembrolizumab) Therapy on Intratumoral Immune Infiltrates in Renal Cell Cancer (RCC) Patients Undergoing Surgical Resection
Brief Title: A Study Evaluating the Effect of Pembrolizumab (MK-3475) in Participants With Renal Cell Cancer (MK-3475-031)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated early due to low enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-031; 2014-002526-12 (EudraCT Number); MK-3475-031 (Other: Merck); KEYNOTE-031 (Other: Merck)
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Results first posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-06

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant Pembrolizumab + RCC Resection (Experimental): Participants received pembrolizumab, 200 mg intravenously (IV) once every 3-week cycle for up to 2 cycles followed by standard of care (SOC) renal cell carcinoma (RCC) surgical resection; and then received post-resection pembrolizumab 200 mg IV once every 3 week cycle for up to approximately 1 year (17 cycles). Post-resection pembrolizumab was only administered to participants who enrolled after Protocol Amendment 04.
  Interventions: Drug: Pembrolizumab Pre-Resection; Procedure: Surgical Resection; Drug: Pembrolizumab Post-Resection
- RCC Resection (Experimental): Participants received SOC renal cell carcinoma (RCC) surgical resection; and then may have received post-resection pembrolizumab 200 mg IV once every 3 week cycle for up to approximately 1 year (17 cycles). Post-resection pembrolizumab was only administered to participants who enrolled under Protocol Amendment 04.
  Interventions: Procedure: Surgical Resection; Drug: Pembrolizumab Post-Resection

INTERVENTIONS:
Drug: Pembrolizumab Pre-Resection — 200 mg administered by IV, once every 3-week cycle for a maximum of 2 cycles
  Other Names: KEYTRUDA®; MK-3475
  Arms: Neoadjuvant Pembrolizumab + RCC Resection
Procedure: Surgical Resection — Standard of care surgical resection of RCC tumor
Drug: Pembrolizumab Post-Resection — 200 mg administered by IV, once every 3-week cycle for a maximum of 17 cycles
  Other Names: KEYTRUDA®; MK-3475

SUMMARY:
This study will examine the effect of treatment with the neoadjuvant antibody pembrolizumab (MK-3475) on tumors of participants with renal cell cancer (RCC). The primary hypotheses are that pembrolizumab is well tolerated in participants undergoing RCC tumor resection; and that pembrolizumab will stimulate a 2-fold or greater increase in intratumoral lymphocytic infiltration in at least 30% of participants with RCC.

ELIGIBILITY:
Inclusion Criteria:

* Have a newly diagnosed RCC, with a primary tumor diameter of more than 4 cm (>= T1b), not previously treated, and be a candidate for operative tumor resection
* Be willing and able to undergo pre-treatment baseline image-guided core biopsy of their primary RCC
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Demonstrate adequate organ function
* Female is not breast feeding, is postmenopausal or surgically sterile; demonstrates non-pregnant state, and agrees to use two acceptable methods of birth control throughout the trial, until 120 days after the last dose of treatment
* Male with female partner of childbearing potential agrees to use adequate method of contraception throughout study, until 120 days after last dose of treatment or last blood draw.

Exclusion Criteria:

* Is currently participating in, or has participated in a study with an investigational agent or device within 4 weeks prior to first dose of study therapy
* Has a diagnosis of immunosuppression or has received systemic steroid therapy, or any other form of immunosuppressive therapy within 4 weeks prior to first dose of study therapy
* Has had prior chemotherapy, targeted small molecule, or radiation therapy for treatment of RCC
* Has a known additional (other than RCC) malignancy that is progressing or requires active treatment
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active, or documented history of autoimmune disease, with the exceptions of vitiligo or resolved childhood asthma/atopy
* Has a history of (non-infectious) pneumonitis that required treatment with steroids or current pneumonitis.
* Has an active infection requiring systematic therapy
* Is receiving anticoagulant therapy, with the exception of low dosage aspirin
* Has severe cardiovascular disease or symptomatic ischemic heart disease
* Has hepatic decompensation
* Has uncontrolled thyroid dysfunction
* Has uncontrolled diabetes mellitus
* Has known psychiatric or substance abuse disorders
* Female is pregnant or breastfeeding
* Is expecting to conceive children within the projected maximum duration of the trial, extending through 120 days after the last dose of treatment or the last blood draw
* Has received prior therapy with any antibody or drug (including ipilimumab) specifically targeting T-cell co-stimulation or checkpoint pathway
* Has a known history of human immunodeficiency virus (HIV)
* Has known active hepatitis B or C
* Has received a live vaccine within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection | RCC Resection
Started | 6 | 4
Received Neoadjuvant Pembrolizumab | 4 | 0
Underwent RCC | 4 | 3
Received Post-RCC Pembrolizumab | 1 | 1
Completed | 4 | 3
Not Completed | 2 | 1
Not completed — Tumor not of the required cell histology | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease progression prior to RCC surgery | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection | RCC Resection | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (5.2) | 55.3 (9.1) | 62.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE) During the Neoadjuvant Pembrolizumab Regimen
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who experienced an AE during their regimen of neoadjuvant pembrolizumab was presented.
Time Frame: Up to Week 16
Population: Per protocol, the analysis population consisted of all participants who received ≥1 dose of neoadjuvant pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an Adverse Event
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who discontinued study drug due to an adverse event is presented.
Time Frame: Up to 56 weeks
Population: The analysis population consisted of all participants who received ≥1 dose of pembrolizumab. Participants in the RCC Resection arm only received pembrolizumab if they enrolled under protocol amendment 04. Counts were based on which course of pembrolizumab (neoadjuvant or post-resection) a participant was receiving at the time of discontinuation.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection | RCC Resection
Number analyzed (Participants) | 4 | 1
Participants
  During neoadjuvant pembrolizumab: number analyzed (Participants) | 4 | 0
  During neoadjuvant pembrolizumab | 0 | 0
  During post-RCC resection pembrolizumab: number analyzed (Participants) | 1 | 1
  During post-RCC resection pembrolizumab | 1 | 0

3. Primary Outcome: Number of Participants Treated With Neoadjuvant Pembrolizumab With a 2-fold or Greater Change From Baseline in Intratumoral CD3+ Lymphocytic Infiltration
Description: The number of participants who received neoadjuvant pembrolizumab and showed a 2-fold or greater change from baseline in intratumoral CD3+ lymphocytic infiltration is presented. Evaluations were based on pathologist score.
Time Frame: Baseline and Week 7
Population: The analysis population consisted of all participants who received ≥1 dose of neoadjuvant pembrolizumab and whose samples were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection
Number analyzed (Participants) | 4
Participants | 1

4. Secondary Outcome: Change From Baseline in Levels of Gene Expression of Immune Modulatory Receptors in Tumors of Participants Treated With Neoadjuvant Pembrolizumab
Description: The change from baseline in levels of gene expression of immune modulatory receptors in tumors of participants treated with neoadjuvant pembrolizumab was presented.
Time Frame: Baseline and Week 7
Population: The analysis population was planned to consist of all participants who received ≥1 dose of neoadjuvant pembrolizumab. Due to low enrollment, there is no data to analyze for this outcome measure and therefore all participants were excluded from analysis.
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection | RCC Resection
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Number of T Cells in Tumors of Participants Treated With Neoadjuvant Pembrolizumab
Description: The change from baseline in number of T cells in tumors of participants treated with neoadjuvant pembrolizumab was presented.
Time Frame: Baseline and Week 7
Population: as for outcome 4
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection | RCC Resection
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Number of Activated T Cells in Peripheral Blood of Participants Treated With Neoadjuvant Pembrolizumab
Description: The change from baseline in the number of activated T cells in peripheral blood of participants treated with neoadjuvant pembrolizumab was presented.
Time Frame: Baseline and Week 7
Population: as for outcome 4
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection | RCC Resection
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Levels of Programmed Cell Death 1 Ligand 1 (PD-L1) Protein in Tumors of Participants Treated With Neoadjuvant Pembrolizumab
Description: The change from baseline in levels of programmed cell death 1 ligand 1 (PD-L1) protein in tumors of participants treated with neoadjuvant pembrolizumab in participants who received neoadjuvant pembrolizumab was presented.
Time Frame: Baseline and Week 7
Population: as for outcome 4
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection | RCC Resection
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Levels of Programmed Cell Death 1 Ligand 2 (PD-L2) Protein in Tumors of Participants Treated With Neoadjuvant Pembrolizumab
Description: The change from baseline in levels of programmed cell death 1 ligand 2 (PD-L2) protein in tumors of participants treated with neoadjuvant pembrolizumab in participants who received neoadjuvant pembrolizumab was presented.
Time Frame: Baseline and Week 7
Population: as for outcome 4
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection | RCC Resection
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Number of Participants Treated With Neoadjuvant Pembrolizumab With a 2-fold or Greater Change From Baseline in Intratumoral CD8+ Lymphocytic Infiltration
Description: The number of participants who received neoadjuvant pembrolizumab and showed a 2-fold or greater change from baseline in intratumoral CD8+ lymphocytic infiltration is presented. Evaluations were based on pathologist score.
Time Frame: Baseline and Week 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection
Number analyzed (Participants) | 4
Participants | 1

10. Primary Outcome: Number of Participants Treated With Neoadjuvant Pembrolizumab With a 2-fold or Greater Change From Baseline in Intratumoral FoxP3+ Lymphocytic Infiltration
Description: The number of participants who received neoadjuvant pembrolizumab and showed a 2-fold or greater change from baseline in intratumoral FoxP3+ (forkhead box protein P3 positive) lymphocytic infiltration is presented. Evaluations were based on pathologist score.
Time Frame: Baseline and Week 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 77 weeks
Description: Adverse events are reported only for participants who received treatment as described in each arm's description. Deaths are reported for all participants who enrolled, regardless of whether they received treatment.
  Per protocol, disease progression of cancer under study was not considered an adverse event (AE) unless it resulted in hospitalization or death.
Groups:
- Neoadjuvant Pembrolizumab + RCC Resection: Participants received pembrolizumab, 200 mg intravenously (IV) once every 3-week cycle for up to 2 cycles followed by standard of care (SOC) renal cell carcinoma (RCC) surgical resection; and then received post-resection pembrolizumab 200 mg IV once every 3 week cycle for up to approximately 1 year (17 cycles). Post-resection pembrolizumab was only administered to participants who enrolled after Protocol Amendment 04. Adverse events in this arm are only counted until 30 days after RCC resection for non-serious adverse events, 90 days for serious adverse events, or until a participant started the post-surgery course of pembrolizumab, whichever occurred first. Deaths are counted from the time of enrollment until a participant started the post-surgery course of pembrolizumab.
- Neoadjuvant Pembrolizumab+Resection+Post-Surgery Pembrolizumab: Participants received pembrolizumab, 200 mg intravenously (IV) once every 3-week cycle for up to 2 cycles followed by standard of care (SOC) renal cell carcinoma (RCC) surgical resection; and then received post-resection pembrolizumab 200 mg IV once every 3 week cycle for up to approximately 1 year (17 cycles). Post-resection pembrolizumab was only administered to participants who enrolled after Protocol Amendment 04. Adverse events and deaths in this arm are only counted after a participant started the post-surgery course of pembrolizumab.
- SOC RCC Resection: Participants received SOC renal cell carcinoma (RCC) surgical resection; and then may have received post-resection pembrolizumab 200 mg IV once every 3 week cycle for up to approximately 1 year (17 cycles). Post-resection pembrolizumab was only administered to participants who enrolled under Protocol Amendment 04. Adverse events in this arm are only counted until 30 days after RCC resection for non-serious adverse events, 90 days for serious adverse events, or until a participant started the post-surgery course of pembrolizumab, whichever occurred first. Deaths are counted from the time of enrollment until a participant started the post-surgery course of pembrolizumab.
- RCC Resection + Post-Resection Pembrolizumab: Participants received SOC renal cell carcinoma (RCC) surgical resection; and then may have received post-resection pembrolizumab 200 mg IV every 3 week cycle for up to approximately 1 year (17 cycles). Post-resection pembrolizumab was only administered to participants who enrolled under Protocol Amendment 04. Adverse events and deaths in this arm are only counted after a participant started the post-surgery course of pembrolizumab.
Arm/Group | Neoadjuvant Pembrolizumab + RCC Resection | Neoadjuvant Pembrolizumab+Resection+Post-Surgery Pembrolizumab | SOC RCC Resection | RCC Resection + Post-Resection Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/1 | 1/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/1 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 1/1 | 0/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Pembrolizumab + RCC Resection (N=4) | Neoadjuvant Pembrolizumab+Resection+Post-Surgery Pembrolizumab (N=1) | SOC RCC Resection (N=3) | RCC Resection + Post-Resection Pembrolizumab (N=1)
Infections and infestations (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Pembrolizumab + RCC Resection (N=4) | Neoadjuvant Pembrolizumab+Resection+Post-Surgery Pembrolizumab (N=1) | SOC RCC Resection (N=3) | RCC Resection + Post-Resection Pembrolizumab (N=1)
Eye disorders (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
General disorders and administration site conditions (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
General disorders and administration site conditions (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
General disorders and administration site conditions (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
General disorders and administration site conditions (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
Investigations (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
Investigations (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
Nervous system disorders (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 1 (1) — Due to the small sample size for this study, we are not disclosing the specific Adverse Event term for this Adverse Event due to patient confidentiality concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT02212730/Prot_SAP_000.pdf